CLINICAL TRIAL: NCT04572633
Title: The HistoSonics System for Treatment of Primary and Metastatic Liver Tumors Using Histotripsy (#HOPE4LIVER US)
Brief Title: The HistoSonics System for Treatment of Primary and Metastatic Liver Tumors Using Histotripsy
Acronym: #HOPE4LIVER US
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP1427
Record Dates: First submitted 2020-09-28; First posted 2020-10-01 (Actual); Results first posted 2024-04-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Liver Neoplasms; Hepatocellular Carcinoma; Liver Metastases
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: This is a single arm, non-randomized prospective trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HistoSonics System (Experimental)
  Interventions: Device: HistoSonics System

INTERVENTIONS:
Device: HistoSonics System — The HistoSonics System (System) is intended for the destruction of liver tissue using histotripsy, a non-thermal, mechanical process using focused ultrasound.
  Other Names: Histotripsy

SUMMARY:
This trial is a single arm, non-randomized prospective trial. The objective of this trial is to evaluate the efficacy and safety of the HistoSonics System for the treatment of primary or metastatic tumors located in the liver. The co-primary safety and efficacy endpoints must be met for the trial to be successful.

DETAILED DESCRIPTION:
This trial is a single arm, non-randomized, multicenter, prospective trial. Following histotripsy treatment of liver tumor(s), subjects will undergo imaging ≤36 hours post-index procedure to determine technical success. Subjects will then be followed for 30 days. Additionally, subjects will be evaluated at 6 months and followed annually for up to five (5) years post-index procedure.

The #HOPE4LIVER US trial required pooling data from #HOPE4LIVER US and #HOPE4LIVER EU/UK (NCT04573881). Subjects were treated with the same intervention (HistoSonics System) using identical protocols tailored to the regulatory requirements for each geography.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. Subject has signed the Ethics Committee (EC) or Institutional Review Board (IRB) approved trial Informed Consent Form (ICF) prior to any trial related tests/procedures and is willing to comply with trial procedures and required follow-up assessments
3. Subject is diagnosed with hepatocellular carcinoma (HCC) or liver metastases (mets) from other primary cancers
4. Subject is able to undergo general anesthesia
5. Subject has a Child-Pugh Score of A or B
6. Subject has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) grade 0-2 at baseline screening
7. Subject meets the following functional criteria, ≤7 days prior to the index-procedure:

   * Liver function: Alanine transaminase (ALT) and Aspartate transaminase (AST) <2.5x upper limit of normal (ULN) and/or bilirubin <2.5 ULN, and
   * Renal function: serum creatinine <2x ULN, and
   * Hematologic function: neutrophil count >1.0 x 10^9/L and platelet >50 x 10^9/L
8. Subject has an International Normalized Ratio (INR) score of <2.0 , ≤7 days prior to the index procedure
9. Subject has not responded to and/or has relapsed and/or is intolerant of other available therapies including locoregional therapies, chemotherapy, immunotherapy and targeted therapies
10. The tumor(s) selected for histotripsy treatment must be ≤3 cm in longest diameter
11. Subject has an adequate acoustic window to visualize targeted tumor(s) using ultrasound imaging
12. Subject has a maximum of three (3) tumors to be treated with histotripsy during the index procedure, regardless of how many tumors the subject has.

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant or nursing (lactating) during the trial period
2. Subject is enrolled in another investigational trial and/or is taking investigational medication and/or has been treated with an investigational device ≤30-days prior to planned index procedure date
3. In the Investigator's opinion, the subject has co-morbid disease(s) or condition(s) that would cause undue risk and preclude safe use of the HistoSonics System
4. Subject has a serum creatinine >2.0 mg/dL or estimated glomerular filtration rate (EGFR) <30, unless on dialysis
5. Subject has major surgical procedure or significant traumatic injury ≤2 weeks prior to the planned index procedure or not fully recovered (CTCAE grade 1 or better) from side effects/complications of such procedure or trauma
6. Subject has not recovered to common terminology criteria for adverse events (CTCAE) grade 1 or better from any adverse effects (except alopecia, fatigue, nausea, vomiting and peripheral neuropathy) related to previous anti-cancer therapy
7. Subject has a history of, or suspected to have, bleeding disorders that are uncorrectable
8. Subject has coagulopathy that is uncorrectable
9. Subject has a planned cancer treatment (e.g. resection, chemotherapy, etc.) after the planned index-procedure date and prior to completion of the 30-day follow-up visit
10. Subject has previous treatment with bevacizumab that has not been discontinued >40 days prior to the planned index-procedure date
11. Subject has planned bevacizumab treatment prior to completion of the 30-day follow-up visit
12. Subject has previous treatments with chemotherapy and/or radiotherapy that has not been discontinued ≥2 weeks prior to the planned index-procedure date and has not recovered (CTCAE grade 1 or better) from related toxicity (except alopecia and peripheral neuropathy)
13. Subject has previous treatment with immunotherapies that has not been discontinued ≥4 weeks prior to the index-procedure and has not recovered from related toxicity (CTCAE grade 1 or better)
14. Subject has a life expectancy less than six (<6) months
15. In the opinion of the Investigator, histotripsy is not a treatment option for the subject
16. Subject has a concurrent condition that, in the investigator's opinion, could jeopardize the safety of the subject or compliance with the protocol
17. Subjects' tumor(s) is not treatable by the System's working ranges (refer to User Manual)
18. Subject has a known sensitivity to contrast media and cannot be adequately pre-medicated
19. Subjects' target tumor(s) has/have had prior locoregional therapy (e.g. ablation, embolization, radiation)
20. Subject is eligible for surgical resection
21. Targeted tumor(s) treatment volume overlaps a non-targeted tumor visible via imaging
22. The targeted tumor(s) is not clearly visible with diagnostic ultrasound and computed tomography (CT) or magnetic resonance (MR) imaging
23. The targeted tumor(s) is located in liver segment 1
24. The Planned Treatment Volume intended to cover the targeted tumor includes or encompasses any portion of the main portal vein, common hepatic duct, common bile duct, gallbladder or stomach/bowel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2027-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Ziemlewicz, MD, Principal Investigator — University of Wisconsin, Madison; Clifford S Cho, MD, Principal Investigator — University of Michigan
Locations (7):
- United States (7):
  - Miami Cancer Institute, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan Hospital, Ann Arbor, Michigan
  - University Hospital - UW Health, Madison, Wisconsin
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mendiratta-Lala M, Wiggermann P, Pech M, Serres-Creixams X, White SB, Davis C, Ahmed O, Parikh ND, Planert M, Thormann M, Xu Z, Collins Z, Narayanan G, Torzilli G, Cho C, Littler P, Wah TM, Solbiati L, Ziemlewicz TJ. The #HOPE4LIVER Single-Arm Pivotal Trial for Histotripsy of Primary and Metastatic Liver Tumors. Radiology. 2024 Sep;312(3):e233051. doi: 10.1148/radiol.233051. PMID 39225612
- [Result] Ziemlewicz TJ, Critchfield JJ, Mendiratta-Lala M, Wiggermann P, Pech M, Serres-Creixams X, Lubner M, Wah TM, Littler P, Davis CR, Narayanan G, White SB, Ahmed O, Collins ZS, Parikh ND, Planert M, Thormann M, Torzilli G, Solbiati LA, Cho CS. The #HOPE4LIVER Single-arm Pivotal Trial for Histotripsy of Primary and Metastatic Liver Tumors: One-year Update of Clinical Outcomes. Ann Surg. 2025 Dec 1;282(6):908-916. doi: 10.1097/SLA.0000000000006720. Epub 2025 Apr 9. PMID 40201962

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As the #HOPE4LIVER EU/UK and #HOPE4LIVER US trials were developed with an identical study design using the same device, the data from all 47 participants enrolled were pooled for analysis. The pooled data contains 23 participants treated in the US and 24 participants treated in Europe. Data from the first 44/47 participants enrolled were analyzed for primary effectiveness and primary safety. Follow-up beyond 30 days is ongoing.
Period: Overall Study
Arm/Group | HistoSonics System
Started | 47
Completed (No participant completed the trial at 30 days. Primary outcomes were analyzed at 30 days. Follow up is ongoing.) | 0
Not Completed | 47
Not completed — Participant in active follow-up at 30 days | 47

BASELINE CHARACTERISTICS:
Arm/Group | HistoSonics System
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White | 45
  Other | 1
Type of tumor [Count of Participants; unit: Participants]
  Hepatocellular carcinoma | 19
  Liver metastasis | 28

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy: Technical Success
Description: Technical success, defined as the treatment volume/treatment dimensions being greater than or equal to the targeted tumor, and with complete tumor coverage, via computed tomography (CT) or magnetic resonance (MR) imaging. [Core Laboratory Adjudicated] Primary efficacy was assessed per tumor with a performance goal of greater than 70%.
  Primary efficacy was assessed after the first forty (40) consecutive evaluable subjects were enrolled. Evaluable subjects had sufficient CT or MR imaging data to allow the independent core laboratory to evaluate technical success.
Time Frame: ≤36 hours post-index procedure
Population: Primary efficacy was assessed after the first forty (40) consecutive evaluable subjects were enrolled. Evaluable subjects had sufficient CT or MR imaging data to allow the independent core laboratory to evaluate technical success.
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: tumors
Arm/Group | HistoSonics System
Number analyzed (Participants) | 40
Number analyzed (tumors) | 44
percentage of tumors | 95.5 [83.72 to 100]
Statistical Analysis 1: Comparison: HistoSonics System; Test type: Other; Wilson Score = 95.5, 95% CI 2-sided [83.72 to 100] — Bootstrap sampling with replacement method to account for potential within-subject lesion correlations. Subject is the bootstrap sampling unit, 1,000,000 iterations for bootstrap resampling, and the bias-corrected and accelerated method was used

2. Primary Outcome: Primary Safety: Procedure-Related Major Complications
Description: Number of index procedure related major complications, including device-related events defined as Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher toxicities observed up to 30-days post index-procedure. [Clinical Events Committee Adjudicated] Primary safety was assessed per participant with a performance goal of less than 25%.
  Primary safety was assessed on all subjects enrolled, after the first forty (40) consecutive subjects evaluable for technical success were enrolled. Evaluable subjects had sufficient CT or MR imaging data to allow the independent core laboratory to evaluate technical success. Enrollment of 44 total subjects was required to assess forty (40) subjects evaluable for technical success.
Time Frame: 30 days post-index procedure
Population: Primary safety was assessed on all subjects enrolled, after the first forty (40) consecutive subjects evaluable for technical success were enrolled. Evaluable subjects had sufficient CT or MR imaging data to allow the independent core laboratory to evaluate technical success. Enrollment of 44 total subjects was required to assess forty (40) subjects evaluable for technical success.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HistoSonics System
Number analyzed (Participants) | 44
percentage of participants | 6.8 [2.35 to 18.23]
Statistical Analysis 1: Comparison: HistoSonics System; Test type: Other; Wilson Score = 6.8, 95% CI 2-sided [2.35 to 18.23]

3. Secondary Outcome: Technical Success
Description: Technical success, defined as the treatment volume/treatment dimensions being greater than or equal to the targeted tumor, and with complete tumor coverage, via computed tomography (CT) or magnetic resonance (MR) imaging. [Core Laboratory Adjudicated]
Time Frame: ≤36 hours post-index procedure
Population: Five tumors had insufficient imaging data for the core laboratory to evaluate technical success.
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: tumors
Arm/Group | HistoSonics System
Number analyzed (Participants) | 43
Number analyzed (tumors) | 47
percentage of tumors | 95.7 [84.78 to 100]

4. Secondary Outcome: Procedure-Related Major Complications
Description: Number of index procedure related major complications, including device-related events defined as Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher toxicities observed up to 30-days post index-procedure. [Clinical Events Committee Adjudicated]
Time Frame: 30 days post-index procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HistoSonics System
Number analyzed (Participants) | 47
percentage of participants | 6.4 [2.19 to 17.16]

5. Secondary Outcome: Secondary Efficacy: Technique Efficacy
Description: Technique efficacy, defined as the lack of a nodular or mass-like area of enhancement within or along the edge of the treatment volume assessed via CT or MR imaging at 30-days post-procedure. [Core Laboratory Adjudicated]
Time Frame: 30 days post-index procedure
Population: Six of the 47 tumors analyzed for technical success had missing or insufficient imaging data for the core laboratory to evaluate technique efficacy.
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: tumors
Arm/Group | HistoSonics System
Number analyzed (Participants) | 38
Number analyzed (tumors) | 41
percentage of tumors | 82.9 [68.29 to 92.50]

6. Secondary Outcome: Secondary Safety: All Adverse Events
Description: Number of adverse events (serious and non-serious) reported within 30 days post-index procedure. [Clinical Events Committee Adjudicated]
Time Frame: 30 days post-index procedure
Measure: Number; unit: adverse events
Arm/Group | HistoSonics System
Number analyzed (Participants) | 47
adverse events | 108

ADVERSE EVENTS:
Time Frame: Enrollment through 30 days
Description: All adverse events were reported starting at the time the participant was enrolled in the trial to the 1-year visit interval or trial exit (whichever comes first). Data collection for adverse events is still ongoing.
Arm/Group | HistoSonics System
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 9/47
Other Adverse Events (participants affected / at risk) | 35/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HistoSonics System (N=47)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1)
Melaena/Melena (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HistoSonics System (N=47)
Abdominal pain (Gastrointestinal disorders) | 11 (11)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Eructation (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 6 (7)
Fatigue (General disorders) | 5 (5)
Pain (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (2)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Discomfort (General disorders) | 1 (1)
Localized oedema (General disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 11 (11)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1)
Post procedural oedema (Injury, poisoning and procedural complications) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Respiratory rate increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Anaemia/Anemia (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hepatic hypoperfusion (Hepatobiliary disorders) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT04572633/Prot_SAP_000.pdf